CLINICAL TRIAL: NCT04458350
Title: Impact of Randomized Digital Promotions of SNAP Fruit and Vegetable Incentive Program on Farmers' Market Patronage and Sales
Brief Title: SNAP Fruit and Vegetable Incentive Program Digital Promotions for Farmers' Markets
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: United States Department of Agriculture (USDA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Parke Wilde, Professor, Tufts University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 102728-00001
Record Dates: First submitted 2020-06-30; First posted 2020-07-07 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Fruit and Vegetable Intake; Healthy Diet; Food Insecurity
Keywords: Supplemental Nutrition Assistance Program; Incentives; Promotions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital Promotions Group (Experimental): Eligible zip codes (n=96) will be randomized using stratified randomization at the state level. The intervention will last 13 weeks (Summer 2020 market season) and consist of receiving digital ads on the Fresh EBT app and Facebook for SNAP fruit and vegetable incentive programs at farmers' markets.
  Interventions: Behavioral: Digital Promotions Group
- Control Group (No Intervention): No intervention administered. Eligible zip codes (n=96) will be randomized using stratified randomization at the state level.

INTERVENTIONS:
Behavioral: Digital Promotions Group — Digital promotions on the Fresh EBT app and Facebook will run for 13 weeks, advertising a SNAP fruit and vegetable incentive at farmers' markets in New England. The intervention will be applied to zip codes randomized to the intervention arm.
  Arms: Digital Promotions Group

SUMMARY:
The purpose of this study is to assess the impact of digital promotions of a Supplemental Nutrition Assistance Program (SNAP) fruit and vegetable incentive program on SNAP participant patronage and sales at farmers' markets. The study will analyze SNAP transactions from zip codes that receive digital promotions compared to zip codes that receive no additional promotions.

DETAILED DESCRIPTION:
Supplemental Nutrition Assistance Program (SNAP) financial incentives for fruits and vegetables (FV) increase FV purchases and consumption with long-term implications for nutrition-related chronic disease. However, many SNAP participants are not aware of these programs, leaving them underutilized. The investigators aim to assess if digital promotions of SNAP incentive programs increase SNAP patronage and sales at farmers' markets. Eligible farmers' markets in the New England Nutrition Incentives Collaborative (NENIC) will receive digital promotions for their SNAP fruit and vegetable incentive programs on the Fresh EBT app and Facebook, randomly assigned to nearby eligible zip codes. Eligible zip codes will be randomized to receive the intervention (digital promotion) or serve as a comparison (no additional promotion) with ads running for 13 weeks (Summer 2020 market season).

ELIGIBILITY:
Inclusion Criteria:

* Farmers' markets in the New England Nutrition Incentives Collaborative (NENIC) are eligible to participate if they were data compliant in Summer 2019 (>90% SNAP transactions reported with zip codes) and have 2 or more nearby, target zip codes.
* Zip codes are eligible if their zip code tabulation area (ZCTA) centroid is within a 7-mile (urban county) or 16-mile (rural county) travel distance of eligible NENIC farmers' market and the zip code has at least 25 active users on the Fresh EBT app

Exclusion Criteria:

* Zip code is not in Connecticut, Maine, New Hampshire, Rhode Island, or Vermont

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251966 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Average number of market SNAP transactions by zip code for Summer 2020 | 13 weeks
  Participating farmers' markets record individual SNAP transactions, including zip code, and upload transaction data to FM Tracks, an online platform for managing farmers' market sales. Average number of SNAP transactions will be computed.

SECONDARY OUTCOMES:
Average market SNAP-related sales by zip code for Summer 2020 | 13 weeks
  Participating farmers' markets record individual SNAP transactions, including zip code, and upload transaction data to FM Tracks, an online platform for managing farmers' market sales. Average SNAP Electronic Benefit sales and incentives distributed (in dollars) will be computed.
Average market new SNAP customers by zip code for Summer 2020 | 13 weeks
  Participating farmers' markets record individual SNAP transactions, including zip code, and upload transaction data to FM Tracks, an online platform for managing farmers' market sales. Average number of new customers will be computed.

CONTACTS AND LOCATIONS:
Locations (1):
- Tufts University Friedman School of Nutrition Science and Policy, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided